CLINICAL TRIAL: NCT05391412
Title: Effect of Prophylactic Fibrinogen Concentrate In Scoliosis Surgery: A Randomized Pilot Study
Brief Title: Effect of Prophylactic Fibrinogen Concentrate In Scoliosis Surgery
Acronym: EFISS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ondrej Hrdy, Principal Investigator, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT0012022
Record Dates: First submitted 2022-05-02; First posted 2022-05-26 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Fibrinogen; Spine Deformity; Coagulopathy, Consumption; Bleeding
Keywords: fibrinogen; scoliosis; coagulopathy
MeSH Terms: conditions — Disseminated Intravascular Coagulation; Hemorrhage; Scoliosis; Hemostatic Disorders | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fibrinogen group (Experimental): The fibrinogen concentrate (20-30mg/kg, max 2g) will be administered in 100ml (Aqua pro injection) intravenously to the patient.
  Interventions: Drug: Fibrinogen Concentrate Human
- Control group (No Intervention): Patients in the control group will not receive any additional medication than standard of care.

INTERVENTIONS:
Drug: Fibrinogen Concentrate Human — Patients in the intervention group will receive single administration of fibrinogen concentrate intravenously at a dose of 20-30 mg/kg (depending on body weight and clinical condition, according to SmPC). The medicinal product will be diluted in a 100 ml infusion bag and administered after induction of anaesthesia prior beginning of surgery. The infusion rate should not exceed approximately 5 ml per minute.
  Other Names: HAEMOCOMPLETTAN P
  Arms: Fibrinogen group

SUMMARY:
EFISS is a prospective, randomized, placebo-controlled trial testing the feasibility, safety and efficacy of prophylactic administration of fibrinogen in paediatric spinal surgery. The study is monocentric and will be conducted in University Hospital Brno, Czech Republic. This is a pilot study in which the primary objective will be to evaluate the feasibility of a clinical trial in 32 selected patients undergoing scoliosis surgery. Participants will be randomized into study groups in a 1:1 allocation ratio and followed up for 28 days after surgery. The expected duration of this clinical trial is 8 months.

DETAILED DESCRIPTION:
Scoliosis is an abnormal lateral curvature of the spine. It is most commonly diagnosed in childhood and early adolescence. Surgical treatment is indicated for severe scoliosis to reduce back pain, neurological symptoms and prevent deterioration of respiratory and cardiovascular function. Scoliosis surgery is often accompanied by a large blood loss and blood transfusion is necessary in 30% to 60% of operated patients. The limited availability, high cost and risk of complications associated with the administration of transfusion products has led to efforts to introduce procedures that aim to reduce the magnitude of blood loss during surgery. Fibrinogen plays an important role in coagulum formation and bleeding arrest. Insufficient fibrinogen levels lead to impaired blood clotting and increased bleeding during major surgery. It has also been shown that patients with higher preoperative fibrinogen levels have less perioperative blood loss. Prophylactic administration of fibrinogen leads to a reduction in blood loss and the number of transfusions administered in some types of procedures. Prophylactic administration of fibrinogen at a dose of 30 mg/kg has been shown to be safe even in paediatric patients. Whether prophylactic fibrinogen administration before scoliosis surgery has an effect on the magnitude of blood loss is unclear. To plan a sufficiently large randomized trial to clarify the effect of prophylactic fibrinogen administration before elective scoliosis surgery on the magnitude of blood loss, and the need for transfusion administration, our team of investigators decided to organize this pilot study.

Prophylactic administration of fibrinogen has been widely described in various indications in recent decades. Among others, it is mainly cardiovascular surgery, where some authors refer the absence of the effect of fibrinogen administration on postoperative bleeding and some even the association with increased allogeneic blood product transfusion. On the contrary, one-hundred sixteen patients undergoing heart surgery with an expected cardiopulmonary bypass were part of the placebo-controlled double-blind study in which fibrinogen concentrate significantly reduced postoperative bleeding with a significant reduction in allogeneic blood products transfusions. Reduction of bleeding after coronary artery bypass graft without signs of postoperative hypercoagulability associated with preoperative infusion of fibrinogen concentrate is descibed. Fibrinogen administration has also been tested in double-blind placebo-controlled clinical trials associated with urologic surgery and gynaecological surgery procedures. Regarding skeletal surgery, the effect of prophylactically administered fibrinogen on postoperative bleeding has also been studied. Intraoperative administration of fibrinogen was successfully used to significantly decrease bleeding and transfusions in 30 children aged 6 months to 17 years undergoing craniosynostosis surgery.

Compared to these results, no differences in blood loss and transfusion requirements were found between treated and placebo groups in younger paediatric patients up to 25 months during craniofacial surgery. Clinical trials directly related to spinal surgery have also been described. This clinical study was performed in 30 adult patients undergoing lumbar surgery, in which 1g of fibrinogen dissolved in distilled water was injected near the surgical incision in the intervention group (n=15). Bleeding during and after surgery in the control group was significantly higher than in the intervention group (P<0.05), and therefore the efficacy of fibrinogen was demonstrated in this indication. Efficacy and safety of preoperatively administrated fibrinogen concentrate (30 mg / kg to 2 g maximum) have also been confirmed in the paediatric population. A total of 102 children (12 - 18 years) with idiopathic scoliosis undergoing surgery were randomized to test and control groups (n=51), where fibrinogen infusion reduced median perioperative bleeding by approximately 155 ml compared to placebo. Fibrinogen administrated in the test group in this case did not reduce the amount of allogeneic blood product transfusion.

The clinical outcome of an individual participant in the prophylactic administration of fibrinogen prior to scoliosis surgery may or may not be improved. If effective, this administration will reduce blood loss during surgery and reduce the need for blood transfusions. In any case, participation in this study will improve knowledge about the prophylactic use of fibrinogen during scoliosis surgery, and all participants in this study will contribute to this socially beneficial knowledge. The same surgical procedure will be used in both study groups as is standard in the surgical treatment of spinal scoliosis. The method is generally well tolerated by patients and does not pose significant risks. The potential risks of participating in the EFISS study may include the rare development of adverse reactions, including fever, allergic and anaphylactic reactions, or thromboembolic events associated with the administration of investigational medicinal product.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for the trial if they meet all of the following criteria:

1. Age < 18 years of age at the time of enrolment
2. Elective scoliosis surgery
3. Signed the relevant informed consent form (more in Chapter 10.1)
4. Sexually active participants (≥ 15 years old) must agree to the use of following methods of contraception for the duration of this clinical trial:

   1. Women - proper use of a highly reliable method of contraception, i.e. combined hormonal contraception (oral, vaginal or transdermal form), gestagen hormonal contraceptives associated with ovulation inhibition (oral or injectable form) or sexual abstinence.
   2. Men - sexual abstinence or the use of an adequate contraceptive method (i.e. condom) in case of sexual intercourse.

Exclusion Criteria:

Subjects will not be eligible for the trial if they meet any of the following criteria:

1. Diagnosed congenital or acquired coagulopathy
2. Use of anticoagulants with the exception of perioperative prophylactic administration of Low molecular weight heparin (LMWH) to prevent venous thromboembolism (VTE)
3. Known hypersensitivity to the active substance or to any of the excipients of Investigational Medicinal Product (IMP)
4. History of deep vein thrombosis or pulmonary embolism
5. Pregnancy and lactation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event | through study completion, an average of 6 months
  The following primary endpoint will be monitored to evaluate the primary objective:
  Adverse event - Any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Adverse drug reaction | through study completion, an average of 6 months
  The following primary endpoint will be monitored to evaluate the primary objective:
  Adverse drug reaction - All untoward and unintended responses to an investigational medicinal product related to any dose administered
Serious adverse event and reaction | through study completion, an average of 6 months
  The following primary endpoint will be monitored to evaluate the primary objective:
  Serious adverse event and reaction - A serious adverse event/reaction is any untoward medical occurrence or effect that at any dose:
  * Results in death;
  * Is life-threatening;
  * Requires hospitalization or extension of existing hospitalization;
  * Results in persistent or significant disability or incapacity;
  * Is a congenital anomaly or birth defect
Unexpected adverse reaction | through study completion, an average of 6 months
  The following primary endpoint will be monitored to evaluate the primary objective:
  Unexpected adverse reaction - Adverse reaction, the nature, severity, or outcome of which
Suspected unexpected serious adverse reaction | through study completion, an average of 6 months
  The following primary endpoint will be monitored to evaluate the primary objective:
  Suspected unexpected serious adverse reaction - Any suspected adverse reaction related to the study treatment that is both serious and unexpected.

SECONDARY OUTCOMES:
Deep-vein thrombosis | through study completion, an average of 6 months
  Incidence of adverse events and reactions according to following Adverse Events of Special Interest (AESI)
  ▪ Deep-vein thrombosis verified on duplex ultrasound imaging (YES/NO)
Pulmonary embolism | through study completion, an average of 6 months
  Incidence of adverse events and reactions according to following Adverse Events of Special Interest (AESI)
  ▪ Pulmonary embolism confirmed on CT (YES/NO)
Infection or healing disorder | through study completion, an average of 6 months
  Incidence of adverse events and reactions according to following Adverse Events of Special Interest (AESI)
  ▪ Infection or healing disorder requiring re-surgery and / or initiation of antibiotic therapy (YES/NO)
Length of stay | through study completion, an average of 6 months
  ▪ Length of stay (LOS) - day of admission - day of discharge will be counted as 1 day
ICU length of stay | through study completion, an average of 6 months
  ▪ ICU length of stay (ICU LOS) - day of admission - day of discharge will be counted as 1 day
28-day mortality | at day 28 of study
  ▪ 28-day mortality (number of patients who are not alive 28 days after randomization)
Age | at the start of the study
  Comparison of demographic characteristics between study groups
  ▪ Age (years)
Sex | at the start of study
  Comparison of demographic characteristics between study groups
  ▪ Sex (male, female)
Weight | at the start of study
  Comparison of demographic characteristics between study groups
  ▪ Weight (kilograms)
Haemoglobin | before surgery, immediately after surgery and 24 hours after surgery
  Comparison of laboratory values of selected haematological parameters between study groups
  ▪ Haemoglobin (g/l; before, at the end of surgery and 24 hours after surgery)
Haematocrit groups | before surgery, immediately after surgery and 24 hours after surgery
  Comparison of laboratory values of selected haematological parameters between study
  ▪ Haematocrit (%; before, at the end of surgery and 24 hours after surgery)
Platelet count | before surgery, immediately after surgery and 24 hours after surgery
  Comparison of laboratory values of selected haematological parameters between study groups
  ▪ Platelet count (n/l; before, at the end of surgery and 24 hours after surgery)
Fibrinogen | before surgery, immediately after surgery and 24 hours after surgery
  Comparison of laboratory values of selected haematological parameters between study groups
  ▪ Fibrinogen (g/l; before, at the end of surgery and 24 hours after surgery)
Activated parcial thromboplastin time (aPTT) | before surgery, immediately after surgery and 24 hours after surgery
  Comparison of laboratory values of selected haematological parameters between study groups
  ▪ aPTT (s; before, at the end of surgery and 24 hours after surgery)
Prothrombin time (PT) | before surgery, immediately after surgery and 24 hours after surgery
  Comparison of laboratory values of selected haematological parameters between study groups
  ▪ PT (s; before, at the end of surgery and 24 hours after surgery)
Thrombin time (TT) | before surgery, immediately after surgery and 24 hours after surgery
  Comparison of laboratory values of selected haematological parameters between study groups
  ▪ TT (s; before, at the end of surgery and 24 hours after surgery)
Total volume of blood loss | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Total volume of blood loss (ml; during surgery and in the 24-hour postoperative period)
Number of the surgical segments of the spine | immediately after surgery
  Comparison of blood loss level and its compensation between study groups
  ▪ Number of the surgical segments of the spine (n; postoperatively)
Volume of blood loss for the surgical segment of the spine | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Volume of blood loss for the surgical segment of the spine (ml; during surgery and in the 24-hour postoperative period)
Urinary output | within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Urinary output (ml; in the 24-hour postoperative period)
Red blood cells (RBC) consumption - transfusion unit | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Red blood cells (RBC) consumption (transfusion units consumption during surgery and in the 24-hour postoperative period)
Red blood cells (RBC) consumption - volume | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Red blood cells (RBC) consumption (total volume of infusion during surgery and in the 24-hour postoperative period)
Thrombocytes of apheresis (TAD) consumption - transfusion unit | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Thrombocytes of apheresis (TAD) consumption (transfusion units consumption during surgery and in the 24-hour postoperative period)
Thrombocytes of apheresis (TAD) consumption - volume | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Thrombocytes of apheresis (TAD) consumption (total volume of infusion during surgery and in the 24-hour postoperative period)
Fresh frozen plasma (FFP) consumption - transfusion unit | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Fresh frozen plasma (FFP) consumption (transfusion units consumption during surgery and in the 24-hour postoperative period)
Fresh frozen plasma (FFP) consumption - volume | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ TFresh frozen plasma (FFP) consumption (total volume of infusion during surgery and in the 24-hour postoperative period)
Fibrinogen concentrate consumption | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Fibrinogen concentrate consumption (consumption in grams during surgery and in the 24-hour postoperative period)
Prothrombin complex concentrate (PCC) consumption | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Prothrombin complex concentrate (PCC) consumption (consumption in units during surgery and in the 24-hour postoperative period)
Blood derivative corresponding to Fresh frozen plasma (Octaplas) consumption | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Blood derivative corresponding to Fresh frozen plasma (Octaplas) consumption (consumption in units during surgery and in the 24-hour postoperative period)
Crystalloid solutions consumption | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Crystalloid solutions consumption (total volume of infusion during surgery and in the 24-hour postoperative period)
Colloid solutions consumption | during surgery and within the 24-hour postoperative period
  Comparison of blood loss level and its compensation between study groups
  ▪ Colloid solutions consumption (total volume of infusion during surgery and in the 24-hour postoperative period)
Number of patients receiving transfusion products | at hospital discharge
  Comparison of blood loss level and its compensation between study groups
  ▪ Number of patients receiving transfusion products
Number of patients receiving blood derivatives | at hospital discharge
  Comparison of blood loss level and its compensation between study groups
  ▪ Number of patients receiving blood derivatives
Rate of recruitment of eligible patients who were approached for consent to participate | through study completion, an average of 6 months
  Feasibility assessment
  ▪ Rate of recruitment of eligible patients who were approached for consent to participate (%; feasibility criterion >75% enrolled participants)
Percentage of missing outcome and clinical data | through study completion, an average of 6 months
  Feasibility assessment
  ▪ Percentage of missing outcome and clinical data (< 10% missing outcome data including ICU and hospital length of stay (LOS) and survival; < 10% missing clinical data obtained from clinical medical notes and electronic patient records)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, M.D., PhD., Principal Investigator — Masaryk University Brno and University Hospital
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hudec J, Vrbica K, Hrdy O, Galko M, Repko M, Stepanova R, Demlova R, Kubelova M, Gal R. Effect of prophylactic fibrinogen concentrate in scoliosis surgery (EFISS): a randomised pilot trial. BMJ Open. 2025 Oct 7;15(10):e100137. doi: 10.1136/bmjopen-2025-100137. PMID 41062134
- [Derived] Vrbica K, Hudec J, Hrdy O, Galko M, Horalkova H, Demlova R, Kubelova M, Repko M, Gal R. Effect of Prophylactic Fibrinogen Concentrate In Scoliosis Surgery (EFISS): a study protocol of two-arm, randomised trial. BMJ Open. 2023 May 26;13(5):e071547. doi: 10.1136/bmjopen-2022-071547. PMID 37236666